CLINICAL TRIAL: NCT07365332
Title: An Adaptive, 2-Part, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of IKT-001 in Pulmonary Arterial Hypertension (PAH)
Brief Title: An Adaptive Program of IKT-001 in Pulmonary Arterial Hypertension (PAH)
Acronym: IMPROVE-PAH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Inhibikase Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IKT-001-201
Record Dates: First submitted 2026-01-22; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: Adaptive, 2-part, randomized, multicenter, double-blind, placebo-controlled, parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IKT-001 (Experimental): IKT-001 tablets for PO administration
  Interventions: Drug: IKT-001
- Placebo (Placebo Comparator): Matching placebo to IKT-001 tablets for PO administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IKT-001 — IKT-001 tablets for PO administration
  Arms: IKT-001
Drug: Placebo — Placebo to IKT-001 tablets for PO administration
  Arms: Placebo

SUMMARY:
This is an adaptive, 2-part, randomized, multicenter, double-blind, placebo-controlled, parallel-group study designed to evaluate the efficacy and safety of IKT-001 in adult participants with WHO Group 1 PAH.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of WHO PAH Group 1 in any of the following subtypes:

  * Idiopathic PAH
  * Heritable PAH
  * Drug/toxin-induced PAH
  * PAH associated with connective tissue disease (CTD)
  * PAH associated with simple, congenital systemic-to-pulmonary shunts at least 1 year following repair
* Men and women 18 and 75 years of age (inclusive)
* Must have a body mass index (BMI) of ≥18.5 kg/m^2 and ≤35.0 kg/m^2 at screening.
* Baseline RHC performed during the Screening Period documenting a PVR of ≥ 400 dyn/sec/cm^5 ; pulmonary capillary wedge pressure (PCWP) ≤15 mmHg and mean pulmonary artery pressure (mPAP) >20 mmHg. PVR enrichment criteria to ensure population baseline PVR >700 dynes/sec/cm^5
* On stable doses of background PAH therapy including endothelin receptor antagonists, phosphodiesterase-5 inhibitors, prostacyclins, and soluble guanylate cyclase stimulators for ≥90 days prior to screening. Current use of sotatercept is not permitted.
* 6MWD ≥ 100 and ≤ 475 m

Exclusion Criteria:

* Diagnosis of PAH WHO Groups 2, 3, 4, or 5.
* Diagnosis of the following PAH Group 1 subtypes: human immunodeficiency virus (HIV)-associated PAH, PAH associated with portal hypertension, schistosomiasis-associated PAH, and pulmonary veno-occlusive disease.
* Any of the following blood pressure-related values or abnormalities: Uncontrolled systemic hypertension as evidenced by sitting systolic BP >160 mmHg or sitting diastolic BP >100 mmHg at screening, Baseline systolic BP <90 mmHg at screening, Syncope within 3 months prior to screening
* History of restrictive, constrictive, or congestive cardiomyopathy.
* ECG with Fridericia's corrected QT interval (QTcF) ≥ 450 msec in males or ≥ 470 msec in females at screening or ≥500 msec in the presence of a right bundle branch block.
* Personal or family history of long QT syndrome or sudden cardiac death.
* Presence of a CardioMEMS device or any other implanted hemodynamic monitoring device.
* Forced vital capacity (FVC) <70 percent on pulmonary function test (PFT) performed no more than 6 months prior to screening; or if FVC is 60 percent to 69 percent, must have a chest computed tomography scan within 12 months with no more than mild interstitial lung disease.
* History of atrial fibrillation or atrial flutter.
* History of cerebrovascular accident, intracranial hemorrhage, or subdural hematoma at anytime, or a fall associated with head trauma within 3 months of screening.
* Acutely decompensated right heart failure within 30 days prior to screening, as per investigator assessment.
* Clinically significant ischemic, valvular, constrictive heart disease, or heart failure with preserved ejection fraction in the opinion of the investigator.
* History of pneumonectomy.
* Untreated or inadequately treated (in the opinion of the investigator) obstructive sleep apnea.
* Acute or chronic hepatitis B or C infection, defined as:

  * Hepatitis B virus: a positive hepatitis B surface antigen test or a positive hepatitis B core antibody test with detectable DNA
  * Hepatitis C virus (HCV): a positive hepatitis C antibody test with detectable HCV ribonucleic acid (RNA).Participants with a positive hepatitis C antibody test, but no detectable HCV RNA who completed treatment with direct-acting antivirals may be considered after discussion with the medical monitor.
* History of or currently diagnosed with a bleeding disorder, including but not limited to hemophilia, von Willebrand disease, thrombocytopenia, or significant bleeding history defined as any bleeding event requiring medical intervention.
* Received treatment with any of the following excluded medications:

  * Currently receiving strong cytochrome P450 (CYP) 3A inducers or CYP3A inhibitors (except for topical administration)
  * Currently receiving or anticipated need to receive any anticoagulant (e.g., heparins, vitamin K antagonists, direct oral anticoagulants, or direct thrombin inhibitors).
  * Current use of sotatercept. Note: participants who previously received sotatercept may be considered if the last dose administered was >6 months prior to screening, participant had no significant bleeding events while on sotatercept.
* Initiation of an exercise program for cardiopulmonary rehabilitation within 90 days prior to screening or planned initiation during the study (participants who are stable in the maintenance phase of a program and who will continue for the duration of the study are eligible).
* History of atrial septostomy within 180 days prior to screening.
* Current participation in another investigational clinical trial and/or receipt of any investigational medication within 90 days prior to screening.
* Previous randomization into this or another IKT-001 study.
* Any social, behavioral, or medical reason that would preclude completion of the study, in the judgement of the investigator.
* Currently lactating, pregnant or planning on becoming pregnant during the study.
* Prior receipt of a solid organ transplant or stem cell transplant.
* Planned surgery that would require any study drug interruption or interfere with study assessments during the study (minor procedures may be allowed in consultation with the medical monitor).
* Malignancy within the last 5 years prior to consent except completely treated non-metastatic-basal cell, squamous cell, in situ cervical cancer, and clinically localized National Comprehensive Cancer Network very low to low risk prostate cancer under active surveillance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
[Part A] To evaluate the effect on Pulmonary Vascular Resistance (PVR) in participants with WHO Group 1 PAH treated with IKT-001 compared to placebo | Baseline to Week 24
  Change in Pulmonary Vascular Resistance (PVR)
[Part B] To characterize the effects of IKT-001 on symptoms and characteristics of Pulmonary Arterial Hypertension compared to placebo | Baseline to Week 24
  Change in 6-minute walk distance (6MWD)

SECONDARY OUTCOMES:
To characterize the effects of IKT-001 on WHO Functional Class | Baseline up to Week 48
  Change in WHO Functional Class
To characterize the effects of IKT-001 on time to clinical worsening | Baseline up to Week 48
  Time to clinical worsening

IPD SHARING:
Plan to Share IPD: No